CLINICAL TRIAL: NCT02332200
Title: Rest Before Physical Therapy in Adolescents With Active Spondylolysis and Spondylolisthesis.
Status: Completed | Type: Observational
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Mitchell Selhorst, Physical Therapist/Research Coordinator, Nationwide Children's Hospital
Other Study IDs: IRB14-00848
Record Dates: First submitted 2015-01-05; First posted 2015-01-06 (Estimated); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Spondylolysis; Spondylolisthesis; Low Back Pain
Keywords: Spondylolysis; Spondylolisthesis; Low Back Pain
MeSH Terms: conditions — Spondylolysis; Spondylolisthesis; Low Back Pain | interventions — Physical Therapy Modalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Early referral to therapy: Patients with a confirmed diagnosis of spondylolysis or spondylolisthesis whose physicians median referral to physical therapy time is less than or equal to 10 weeks.
  Interventions: Other: Physical Therapy
- Later referral to therapy: Patients with a confirmed diagnosis of spondylolysis or spondylolisthesis whose physicians median referral to physical therapy time is >10 weeks.
  Interventions: Other: Physical Therapy

INTERVENTIONS:
Other: Physical Therapy — Physical therapy will consist of standard physical therapy care for spondylolysis or spondylolisthesis.

SUMMARY:
This is a retrospective chart review with a short follow-up phone questionnaire for our patients who have been treated by Nationwide Children's Hospital physical therapy and sports medicine for a spondylolysis or spondylolisthesis injury.

Currently, no research exists to guide referral for safe physical therapy rehabilitation for patients with spondylolysis and spondylolisthesis injuries. By performing this retrospective study the investigators can gain information to better guide physical therapy referral time. This may also serve as foundation for a future prospective randomized trial.

Currently, Nationwide Children Hospital physicians vary from immediate referral to physical therapy to 3 + months of rest prior to beginning therapy. By performing a retrospective chart review assessing time to referral to therapy and patient outcomes the investigator can gain some guidance for when it is safe to prescribe physical therapy rehabilitation for patients with spondylolysis and spondylolisthesis injuries.

Patients with an active spondylolysis or spondylolisthesis injury who are referred to physical therapy early will return to activity/sport sooner without increased risk of adverse reaction.

DETAILED DESCRIPTION:
Spondylolysis is as stress fracture in the pars interarticularis of the vertebral arch most commonly occurring in the lower lumbar spine. Spondylolisthesis is the forward displacement of a vertebra, especially the fifth lumbar vertebra, most commonly occurring after a break or fracture. These injuries to the spine are extremely common in adolescent athletes and some research reports that spondylolysis and spondylolisthesis account for over 40% of all adolescent athletes' low back pain.

While these injuries are common in the adolescent population there is very little research to guide treatment of these patients, particularly with rehabilitation. Conservative standard of care with the treatment of spondylolysis and spondylolisthesis injuries are to rest from sport, brace the lumbar spine, and begin physical therapy and return to sport as the patient is able. There is some evidence to show that patients should rest for 12 weeks prior to returning to sport, otherwise there is an increased risk of injury (El Rassi, 2013). There currently is no research to suggest when to begin physical therapy. Physical therapy for rehabilitation and return to sport is a part of standard of care, but recommendations for beginning therapy vary widely and are not supported by evidence. A concern for beginning physical therapy too soon is that the fracture will not have adequate time to heal and re-injury can occur. While a concern for waiting too long to begin therapy is increased muscle atrophy, high fear avoidance beliefs, and unnecessarily long avoidance of activity.

Currently, Nationwide Children Hospital physician's vary from immediate referral to physical therapy to 3 + months of rest prior to beginning therapy. By performing a retrospective chart review assessing time to referral to therapy and patient outcomes we can gain some guidance for when it is safe to prescribe physical therapy rehabilitation for patients with spondylolysis and spondylolisthesis injuries.

Currently, no research exists to guide referral for safe physical therapy rehabilitation for patients with spondylolysis and spondylolisthesis injuries. By performing this retrospective study we can gain information to better guide physical therapy referral time. This may also serve as foundation for a future prospective randomized trial.

The are two primary objectives of this study: (1) Does time to referral to physical therapy affect time to full return to activity. (2) To assess the safety of an early referral to therapy compared with a long rest period prior to therapy. Safety will be determined by relative risk of adverse reaction and percent of patients able to fully return to activity.

Secondary objectives include:

Assessing pain with early and later referral to therapy. Number of physician visits Number of physical therapy visits Compliance

We will perform a chart review of all spondylolysis and spondylolisthesis patients who have been treated by Nationwide Children's Hospital Sports Medicine physicians and physical therapists since 12/2009 when electronic charting on these patients began. As we are unable to track the outcomes for this study of those patients referred to outside physical therapy, they will be excluded from the study.

The chart review will begin by running a report for all patients with a spondylolysis or spondylolisthesis diagnosis from 2009 to 2013.

Variables that will be automatically pulled in the report will be:

Age at time of diagnosis Gender Treating physician Pain Compliance Sports Played **Any missing variable from the report will be gathered by reviewing the patients chart.** Variables that will be gathered from reviewing the patients chart Diagnosis Level of injury Type of imaging Brace Results of imaging Rest before Physical Therapy Rest before cleared for return to sport Treating physical therapist Number of physical therapy visits Number of physician visits

Variables that will be gathered in a short follow-up survey by contacting the patients. Patients will be contacted by phone, or mail.

Recurrence of symptoms Michelli Function Score Modified Odom's criteria Current level of sport participation

Patients will be divided into 2 groups: Early referral to therapy and late referral to therapy by physician. To account for the fact that patients who are referred to physical therapy sooner may have a less severe injury we will be sub-grouping patients by physician. Patients of a physician with a median referral rate < 10 weeks to therapy will be sub-grouped into Early referral to therapy and patients of a physician with a median referral time >10 weeks will be sub-grouped into Late referral to therapy. To account for possible changes in the way a particular physician treats their patients with a spondylolysis or spondylolisthesis physician referral rate will be assessed yearly and patient grouped based on that calendar year referral rate. For example if a doctor has a median referral rate of 12 weeks to therapy in 2009, but 9 weeks in 2010, their 2010 patients will be placed into the late referral to therapy while there 2010 patients will be placed into the early referral group.

Data Analysis To assess the first primary object we will assess if there is a between group difference (early vs late referral to PT) for time to return sport. We will assess between group differences using a t-test if the data are parametric and a Mann-Whitney U test if the data are nonparametric.

To assess the safety of an early referral to therapy compared with a long rest period prior to therapy. We will examine the relative risk between groups for experiencing a significant recurrence of symptoms.

Secondary Outcomes for the following variables will be assessed by t-test (parametric) or Mann-Whitney U (nonparametric) for continuous data and chi-square analysis for categorical data.

Pain

* PT visits
* physician visits Michelli Function Score Compliance

Descriptive statistics will be reported for all other variables

ELIGIBILITY:
Inclusion Criteria:

* Patient must have been treated by the Nationwide Children's sports medicine physicians as well as Nationwide Children's sports and orthopedic physical therapists for spondylolysis or spondylolisthesis from 2009-2013 confirmed by MRI or Bone Scan.

Exclusion Criteria:

* Diagnosis made by: X-ray, CT, suspicion

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a confirmed diagnosis of spondylolysis and spondylolisthesis who have been treated by Nationwide Children's Hospital Sports Medicine physicians and physical therapists from 12/2009-12/2013.
Sampling Method: Non-Probability Sample
Enrollment: 196 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Rest before cleared for return to sport | Time to event (up to 52 weeks)
  Number of days the patient is at rest per doctor's orders prior to time to return sport. Return to sport is decided by physician's Activity Recommendation for full return to participation. If the physician requests modified participation in their last note, return to sport will be decided by Physical therapist notes. If no mention of full return to sport is made by the physical therapist then the last day of physical therapy will be considered the day the patient made a full return to sport. (This is when the PT decided no more limitations exist)
Significant recurrence of symptoms | At follow-up questionnaire (1-5 years after treatment)
  An unplanned visit to physician due to a worsening of symptom during the treatment of spondylolysis or spondylolisthesis. As well as responding yes to having a significant recurrence reported on follow up questionnaire .

SECONDARY OUTCOMES:
Numeric Pain Rating Scale (NRPS) | Baseline, visit physician prescribes therapy (average 10 weeks after baseline), discharge (average 4-6 month after baseline), and on follow-up questionnaire (1-5 years post treatment)
  Average of the recorded values for NRPS: pain at rest, pain with ADL's, and pain with activity. If the patient is not allowed to participate in activity, pain will be an average of pain at rest and with ADL's.
Number of Physician Visits | Time to discharge from physicians care (up to 104 weeks)
  The number of attended physicians visits for the initial episode of care for treatment of the low back injury only.
Number of Physical Therapy Visits | Time to discharge from physical therapy care (up to 104 weeks)
  The number of attended physical therapy visits for the initial episode of care for treatment of the low back injury only. Physical therapy visits for low back pain prior to rest from sport will be excluded from visit count.
Compliance with prescribed care | Time to discharge from physicians care (up to 104 weeks)
  Reported compliance with physician instructions for care as reported in physician note, if physician makes no comment and the patient attends at least 80% of prescribed physical therapy and physician appointments in the prescribed time frame patient will be considered compliant. (ie 12 physical therapy visits ordered over 6 weeks. Patient must attend 10 visits in 6 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Selhorst, DPT, Principal Investigator — Nationwide Childrens Hospital
Locations (4):
- United States (4):
  - Nationwide Children's Hospital Sports and Ortho PT Ortho Center, Columbus, Ohio
  - Nationwide Children's Hospital Sports and Ortho PT East Broad, Columbus, Ohio
  - Nationwide Children's Hospital Sports and Ortho PT Dublin, Dublin, Ohio
  - Nationwide Children's Hospital Sports and Ortho PT Westerville, Westerville, Ohio

REFERENCES:
- [Derived] Selhorst M, Fernandez-Fernandez A, Schmitt L, Hoehn J. Effect of a Psychologically Informed Intervention to Treat Adolescents With Patellofemoral Pain: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2021 Jul;102(7):1267-1273. doi: 10.1016/j.apmr.2021.03.016. Epub 2021 Apr 7. PMID 33838141
- [Derived] Selhorst M, Fischer A, Graft K, Ravindran R, Peters E, Rodenberg R, MacDonald J. Long-Term Clinical Outcomes and Factors That Predict Poor Prognosis in Athletes After a Diagnosis of Acute Spondylolysis: A Retrospective Review With Telephone Follow-up. J Orthop Sports Phys Ther. 2016 Dec;46(12):1029-1036. doi: 10.2519/jospt.2016.7028. Epub 2016 Nov 8. PMID 27825292